CLINICAL TRIAL: NCT01050751
Title: Open-Label, Randomized, 2-Way Crossover Study To Estimate The Pharmacokinetics And Bioavailability Of Lersivirine (UK 453,061) Administered As A Single 750 Mg Tablet And 3 X 250 Mg Tablets In Healthy Subjects
Brief Title: Bioavailability Of Lersivirine Single 750 Mg Tablet Versus 3 X 250 Mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5271039
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability; Bioequivalence; Lersivirine; UK-453; 061; Pharmacokinetics
MeSH Terms: interventions — UK 453,061

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lersivirine (new formulation) (Experimental)
  Interventions: Drug: Lersivirine
- Lersivirine (old formulation) (Active Comparator)
  Interventions: Drug: Lersivirine

INTERVENTIONS:
Drug: Lersivirine — Oral Lersivirine 750 mg (1 x 750 mg) single dose
  Arms: Lersivirine (new formulation)
Drug: Lersivirine — Oral Lersivirine 750 mg (3 x 250 mg) single dose
  Arms: Lersivirine (old formulation)

SUMMARY:
This is a randomized study to assess whether the pharmacokinetics of a new single 750 mg tablet is similar to 3 x 250 mg tablets (750 mg total).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Treatment with an investigational drug within 30 days or 5 half-lives or local regulation (whichever is longer) preceding the first dose of study medication.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of regular alcohol consumption exceeding 14 drinks/week for women and 21 drinks/week for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To estimate the bioavailability of 1 x 750 mg lersivirine tablet compared to 3 x 250 mg lersivirine tablets. | 7 days

SECONDARY OUTCOMES:
To investigate the safety and tolerability of both single oral 750 mg (3 x 250 mg and 1 x 750 mg) dose of lersivirine. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271039&StudyName=Bioavailability%20Of%20Lersivirine%20Single%20750%20Mg%20Tablet%20Versus%203%20X%20250%20Mg%20Tablets